CLINICAL TRIAL: NCT06855212
Title: A Phase II Study of Neoadjuvant Cetuximab and Cemiplimab in Patients Undergoing Surgery for Head and Neck Squamous Cell Carcinoma
Brief Title: Phase II Study of Neoadjuvant Cetuximab and Cemiplimab in Patients Undergoing Surgery for HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Eli Lilly and Company (Industry); Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23204
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — cemiplimab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Cetuximab and Cemiplimab Treatment (Experimental): Cemiplimab: 350 mg IV dose on C1D1 and C2D1
  Cetuximab: 400mg/m2 loading dose on C1D1 followed by 250 mg/m2 IV weekly doses on C1D8, C1D15, and C2D1 (total 4 doses including the loading dose).
  Interventions: Drug: Cemiplimab; Drug: Cetuximab

INTERVENTIONS:
Drug: Cemiplimab — Given by IV infusion.
Drug: Cetuximab — Given by IV infusion.

SUMMARY:
The purpose of the study is to determine if cemiplimab in combination with cetuximab given before their surgery are beneficial and safe in participants with head and neck squamous cell carcinoma (HNSCC).

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 18 years of age at the time of consent.
* Patient (or a legally authorized representative) must understand and voluntarily sign informed consent prior to any study-related assessments/procedures being conducted.
* Must be able and willing to comply to the study visit schedule and protocol requirements.
* Must have sufficient archived tumor tissue available for PD-L1 CPS determination. If not, patient must agree to a fresh tumor biopsy before starting the treatments. If patient only had a fine needle aspiration, a fresh biopsy with a core needle or punch biopsy is required.
* If the primary site is oropharynx, p16/HPV status must be determined. HPV status determined by cell free HPV DNA testing is also acceptable.
* Must have surgically resectable HNSCC including oral cavity, oropharynx, larynx, and hypopharynx. Patients with p16-positive or HPV-positive unknown primary of head and neck are eligible. Must be newly diagnosed HNSCC with T1-2 N1-3 or T3-4 N0-3 undergoing surgery as a standard of care. If the tumor invades lateral pterygoid muscle, pterygoid plates, lateral nasopharynx, skull base or encases carotid artery, and/or prevertebral fascia involvement, it will be considered as unresectable and excluded.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Must meet the laboratory criteria outlined in the protocol.
* Patients of childbearing potential and patients whose sexual partners are of childbearing potential must be willing to practice an approved method of highly effective birth control with their partners starting at the time of informed consent and for 1 year after the completion of the study treatment regimen. Women of childbearing potential must have a negative pregnancy test within the 7 days prior to enrollment.

Exclusion Criteria:

* Patients with an active autoimmune disease that has required systemic treatment in past 2 years.
* Patients with a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Patient with a history of allergic reactions attributed to compounds of chemical or biologic composition similar to those of cetuximab or if the patient had red meat allergy/tick bite history.
* Patients with an active infection requiring systemic therapy.
* Patients with a known history of human immunodeficiency virus (HIV) infection.
* Patients with a known history of or is positive for Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C (defined as Hepatitis C virus [HCV] ribonucleic acid is detected).
* Patients who have a history of a left ventricular ejection fraction (LVEF) of < 45% or who are New York Heart Association (NYHA) Class 2 or higher.
* Patients with cardiovascular disease defined as: Uncontrolled hypertension defined as blood pressure > 160/90 mmHg at Screening confirmed by repeat (medication permitted). History of torsades de pointes, significant electrocardiogram (ECG) abnormalities, including ventricular rhythm disturbances, unstable cardiac arrhythmia requiring medication, pathologic symptomatic bradycardia, left bundle branch block, second degree atrioventricular (AV) block type II, third degree AV block, Grade ≥ 2 bradycardia, uncorrected hypokalemia not amenable to correction, congenital long QT syndrome, prolonged QT interval due to medications, corrected QT (QTc) > 450 msec (for men) or > 470 msec (for women). Symptomatic heart failure (per New York Heart Association guidelines; (Caraballo, 2019), unstable angina, myocardial infarction, severe cardiovascular disease (ejection fraction < 20%, transient ischemic attack, or cerebrovascular accident within 12 months of Day 1).
* Patients who are of the following protected classes will be excluded: Pregnant, parturient, or breastfeeding women. Persons who are hospitalized without consent because of a judiciary or administrative decision. Patients with a legal protection measure or a person who cannot express his/her consent. Patients in emergency situations who cannot consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Major and Complete Pathologic Response Rate | Day of Surgery
  The number of participants who achieve major or complete pathologic response rate.

SECONDARY OUTCOMES:
Event Free Survival | Up to 24 months
  Event free survival is defined as time from Cycle 1 Day 1 of cetuximab and cemiplimab until disease progression, surgery delayed > 4 weeks from the planned surgery date due to a drug related AE, discontinuation of the neoadjuvant therapy due to a drug related AE, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chung, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States